CLINICAL TRIAL: NCT03466450
Title: Phase Ib/II Multicentric Study Combining Glasdegib (PF-04449913) With Temozolomide in Patients With Newly Diagnosed Glioblastoma, Safety and Preliminary Efficacy for the Combination
Brief Title: Glasdegib (PF-04449913) With Temozolomide Newly Diagnosed Glioblastoma
Acronym: GEINOGLAS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Grupo Español de Investigación en Neurooncología (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GEINO-1602; 2017-002410-31 (EudraCT Number)
Record Dates: First submitted 2018-02-27; First posted 2018-03-15 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Glioblastoma
Keywords: glioblastoma; glasdegib; temozolomide; combined therapy
MeSH Terms: conditions — Glioblastoma | interventions — glasdegib; Temozolomide

STUDY DESIGN:
Intervention Model Description: Phase Ib/II, multicentric, non-randomized, open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Glasdegib and Temozolomide Oral Capsule (Experimental): During Phase Ib, Four to six weeks after surgical diagnosis, concurrent with radiotherapy (STUPP) + temozolomide (75mg/m2/day for 42 days) + PF-04449913 (Glasdegib) (3 dose levels will be evaluated: 100mg QD, 150mg QD and 200mg QD, or 75-50mg) will be administered.
  During Phase II, Radiation therapy, temozolomide and glasdegib will be administered. This last, as the dose that have been selected previously, based on the Phase Ib results. Glasdegib ( PF-04449913) recommended dose until progresion of disease, unacceptable toxicity, non-compliance, consent withdrawal up to 2 years.
  Interventions: Drug: PF-04449913; Drug: Temozolomide Oral Capsule

INTERVENTIONS:
Drug: PF-04449913 — Glasdegib (3 dose levels will be evaluated: 100mg QD, 150mg QD and 200mg QD, or 75-50mg) will be administered:
  During concurrent phase concomitantly with radiation and Extended to the resting period (glasdegib will not be stopped in the 4 weeks of radiotherapy resting period).
  During adjuvant therapy with Temozolomide Oral Capsule. Additional treatment with glasdegib beyond 6 sequential TMZ cycles will continue until progression, unacceptable toxicity, non-compliance, consent withdrawal and/or 2 years of glasdegib administration.
  Other Names: Glasdegib
Drug: Temozolomide Oral Capsule — During RT, patients will receive Temozolamide (TMZ). All patients will be given TMZ at 75 mg/m2
  /d concurrently with RT for a maximum of 42 days. At 4 weeks after RT completion, patients will start taking TMZ at 150 mg/m2/d for the first 5 days of a 28-day cycle. If first cycle is well tolerated, patients will receive TMZ at 200 mg/m2/d for the first 5 days of every subsequent 28-day cycle for another 5 cycles.

SUMMARY:
Glioblastomas (GBMs) are the most common malignant primary brain tumors. Despite multimodality aggressive therapies (surgery followed by chemoradiotherapy based on TMZ and adjuvant TMZ), median overall survival is only 12 to 15 months. This dramatic behavior is mainly due to the high invasiveness and proliferation rate of GBM.

In addition, GBM exhibits a high resistance to standard chemotherapy and radiotherapy. Current strategies for the treatment of GBM are only palliative, and include surgical resection (which is frequently incomplete due to the proximity of the tumour to vital brain structures) and focal radiotherapy. A large number of chemotherapeutic agents (e.g. alkylating agents such as TMZ and nitrosoureas such as carmustine) have also been tested, but they display limited efficacy.

The current gold standard first line treatment for glioma for patients less than 70 years old includes radiation and concurrent TMZ followed by adjuvant TMZ (i.e., the "Stupp regimen"). However, results are disappointing and there is an unmet medical need of new drugs in this setting.

Glasdegib (SHH pathway inhibitor) is a rational therapeutic agent for patients with newly diagnosed Glioblastoma since inhibits SHH pathway interfering with cancer stem cells and endothelial migration.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document.
* Male or Female ≥18 years old.
* Newly diagnosed GBM confirmed by biopsy or resection no more than 4 to 6 weeks before registration.
* Patients candidates for Stupp treatment
* Patients must have at least 15 unstained slides or 1 tissue block (frozen or paraffin embedded) available from a prior biopsy or surgery (archival tumor material).
* Patients must have sufficient time for recovery from prior surgery (at least 4 weeks).
* ECOG ≤ 1.
* Adequate hematologic function: Hematocrit ≥ 29%, Leukocytes > 3,000/mcL, ANC ≥ 1,500 cells/ul, platelets ≥ 100,000 cells/ul.
* Adequate liver function: Bilirubin ≤ 2 x ULN; AST (SGOT) ≤ 2.5 X ULN
* Creatinine within normal institutional limits or creatinine clearance > 60 mL/min for subjects with creatinine levels above institutional normal.
* The effects of SHH pathway inhibitors on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence; surgical sterilization) prior to study entry and for the duration of study participation and for at least 3 months thereafter. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate.

Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. All female patients with reproductive potential must have a negative pregnancy test (serum/urine) within 2 weeks prior to starting treatment.

* Female subjects must either be of non-reproductive potential (ie, post-menopausal by history: ≥60 years old and no menses for ≥1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry.

Exclusion Criteria:

* Presence of extracranial metastatic disease.
* Participants may not be receiving any other investigational agents.
* Patients must not have received prior Gliadel wafers.
* Any surgery (not including minor diagnostic procedures such as lymph node biopsy) within 2 weeks of baseline disease assessments; or not fully recovered from any side effects of previous procedures.
* Any psychiatric or cognitive disorder that would limit the understanding or rendering of informed consent and/or compromise compliance with the requirements of this protocol.
* Any clinically significant gastrointestinal abnormalities, which may impair intake, transit or absorption of the study drug, such as the inability to take oral medication in tablet form.
* Congenital or known history of long QT syndrome, Torsades de pointes, arrhythmias (including sustained ventricular tachyarrhythmia, right or left bundle branch block and bifascicular block, unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure (CHF New York Association class III or IV).
* Current (or within 6 months) significant cardiovascular disease, including, but not limited to myocardial infarction, cerebrovascular accident, transient ischemic attack or symptomatic pulmonary embolism, bradycardia defined as <50 bpms.
* Active cardiac dysrhythmias of NCI CTCAE Grade ≥2 (eg, atrial fibrillation) or QTcF interval (QTc using Fridericia's formula) >470 msec.
* Active and clinically significant infections.
* Current use or anticipated requirement for drugs known to be moderate or strong cytochrome p450 inhibitors.
* Individuals with a history of a different malignancy are ineligible except for the following circumstances: Individuals with a history of other malignancies are eligible if they have been disease-free for at least 3 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 3 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.

Patients will not be eligible if they have evidence of other malignancy requiring therapy other than surgery within the last 3 years.

* Patients who have had prior stereotactic radiotherapy, convection enhanced delivery or brachytherapy (as gliosis/scarring from these modalities may limit delivery).
* Patients will not be eligible if they present with leptomeningeal dissemination.
* Pregnant women are excluded from this study because the potential for teratogenic or abortifacient effects is unknown (glasdegib has been shown to be teratogenic in nonclinical embryo-fetal development studies in rats and mice at subtherapeutic exposures). Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother, breastfeeding should be discontinued if the mother is treated.
* HIV-positive individuals on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions. In addition, these individuals are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to glasdegib.
* Other severe acute or chronic medical condition, uncontrolled intercurrent illness or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgment of the investigator, would make the patient inappropriate for entry into this trial.
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ highly effective birth control from screening to 180 days after the last dose of the study treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
Glasdegib Dose | 12 weeks
  For Phase Ib, The recommended dose for phase 2 (RDP2) of Glasdegib administered with temozolomide during and after RT.
Overall survival | 15 months
  For Phase II, time between the start of treatment to death

SECONDARY OUTCOMES:
Progression Free Survival | 24 months
  Time between the start of treatment and progression of disease
Adverse events (safety) | 24 months
  Based on the number and type of adverse events reported since the start of treatment and throughout the study period.
Response to treatment | 24 months
  Based on RANO criteria

CONTACTS AND LOCATIONS:
Overall Officials: María Angeles Vaz, M.D., Study Chair — Hospital Universitario Ramón y Cajal
Locations (8):
- Spain (8):
  - Institut Catalá de Oncología Badalona/Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Institut Catalá de Oncología Girona/Hospital Universitari Dr. Josep Trueta, Girona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario y Politécnico La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No